CLINICAL TRIAL: NCT01581008
Title: Implementing Collaborative Care to Alleviate Symptoms and Adjust to Heart Failure: A Pilot Study
Brief Title: Improving Symptoms and Quality of Life in Chronic Heart Failure: Pilot Study
Acronym: CASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RRP 11-239; CRICC Pilot (Other Grant/Funding Number: Denver REAP (CRICC) Pilot Grant)
Record Dates: First submitted 2011-10-31; First posted 2012-04-19 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: palliative care; heart failure; delivery of health care
MeSH Terms: conditions — Heart Failure | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Care to Alleviate Symptoms and Adjust to Illness (Experimental): A palliative symptom management and psychosocial care intervention named Collaborative Care to Alleviate Symptoms and Adjust to Illness (CASA) that includes (a) evidence-based palliative symptom management of breathlessness, fatigue, and pain, provided by a nurse; (b) a 6-session structured psychosocial care protocol targeting depression and adjustment to illness, supplemented by informal (family) caregiver assessment and support, provided by a social worker or psychologist; and (c) brief weekly team meetings with the nurse, social worker/psychologist and a palliative care specialist, cardiologist, and primary care provider.
  Interventions: Other: Collaborative Care to Alleviate Symptoms and Adjust to Illness
- Psychospiritual (Active Comparator): A psychospiritual intervention that is home-based, self-guided, and requires minimal resources. It will be delivered in written modular form via US Mail along with brief weekly telephone support.
  Interventions: Behavioral: Psychospiritual

INTERVENTIONS:
Other: Collaborative Care to Alleviate Symptoms and Adjust to Illness — A palliative symptom management and psychosocial care intervention named Collaborative Care to Alleviate Symptoms and Adjust to Illness (CASA) that includes (a) evidence-based palliative symptom management of breathlessness, fatigue, and pain, provided by a nurse; (b) a 6-session structured psychosocial care protocol targeting depression and adjustment to illness, supplemented by informal (family) caregiver assessment and support, provided by a social worker or psychologist; and (c) brief weekly team meetings with the nurse, social worker/psychologist and a palliative care specialist, cardiologist, and primary care provider.
  Other Names: Palliative symptom management and psychosocial care
  Arms: Collaborative Care to Alleviate Symptoms and Adjust to Illness
Behavioral: Psychospiritual — A psychospiritual intervention that is home-based, self-guided, and requires minimal resources. It will be delivered in written modular form via US Mail along with brief weekly telephone support.
  Arms: Psychospiritual

SUMMARY:
The overall goal of this study is to evaluate the pilot implementation of two palliative care interventions in veterans with chronic heart failure at the Denver VA Medical Center. This is a study of behavioral and care strategy interventions and involves no investigational drugs or devices.

DETAILED DESCRIPTION:
The investigators will examine the feasibility of two palliative care interventions designed to improve different facets of quality of life. Briefly, the two interventions are:

1. A palliative symptom management and psychosocial care intervention named Collaborative Care to Alleviate Symptoms and Adjust to Illness (CASA) that includes

   1. evidence-based palliative symptom management of breathlessness, fatigue, and pain, provided by a nurse;
   2. a 6-session structured psychosocial care protocol targeting depression and adjustment to illness, supplemented by informal (family) caregiver assessment and support, provided by a social worker or psychologist; and
   3. brief weekly team meetings with the nurse, social worker/psychologist and a palliative care specialist, cardiologist, and primary care provider.
2. A psychospiritual intervention that is home-based, self-guided, and requires minimal resources. It will be delivered in written modular form via US Mail along with brief weekly telephone support.

The specific aims of the study are to:

1. Examine intervention feasibility and determine preliminary estimates of intervention effect

   1. Determine patient participation rates and cohort retention
   2. Conduct a preliminary assessment of outcomes by measuring pre-post changes in quality of life, depressive symptoms, health status, life meaning, and spirituality.
2. Obtain qualitative feedback from study participants, the persons providing the intervention, and providers/leaders in primary care, mental health, palliative care, chaplaincy, and hospital operations.

ELIGIBILITY:
Inclusion Criteria:

* eligible veterans from the Denver VAMC will have a prior primary discharge diagnosis of heart failure in the last year,
* be at least 18 years of age, able to read and understand English,
* have consistent access to a telephone
* at least one of the following:

  1. Kansas City Cardiomyopathy Questionnaire (KCCQ) score less than or equal to 60;
  2. a second hospitalization for with a primary discharge diagnosis of heart failure in the last year;
  3. taking at least 80 mg oral furosemide (or equivalent) daily in a single or divided dose for at least 2 weeks;
  4. BNP greater than or equal to 250 or NT-proBNP greater than or equal to 1000; or
  5. estimated creatinine clearance 30-80 mL/min.

Exclusion Criteria:

* previous diagnosis of dementia;
* active substance abuse, defined as an AUDIT-C score greater than 7, two positive responses on substance abuse screening questions, or medical records indicating active substance abuse or dependence;
* comorbid metastatic cancer, given the focus on heart failure palliative care;
* nursing home resident; and
* diagnosis of bipolar disorder or schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bekelman, MD MPH, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado, United States

REFERENCES:
- [Result] Bekelman DB, Hooker S, Nowels CT, Main DS, Meek P, McBryde C, Hattler B, Lorenz KA, Heidenreich PA. Feasibility and acceptability of a collaborative care intervention to improve symptoms and quality of life in chronic heart failure: mixed methods pilot trial. J Palliat Med. 2014 Feb;17(2):145-51. doi: 10.1089/jpm.2013.0143. Epub 2013 Dec 11. PMID 24329424
- [Result] Hooker SA, Ross K, Masters KS, Park CL, Hale AE, Allen LA, Bekelman DB. Denver Spirited Heart: Mixed-Methods Pilot Study of a Psychospiritual Intervention for Heart Failure Patients. J Cardiovasc Nurs. 2017 May/Jun;32(3):226-235. doi: 10.1097/JCN.0000000000000337. PMID 27076391

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was a screen failure, thus 30 patients completed baseline surveys and were randomized.
Groups:
- CASA: A palliative symptom management and psychosocial care intervention named Collaborative Care to Alleviate Symptoms and Adjust to Illness (CASA) that includes (a) evidence-based palliative symptom management of breathlessness, fatigue, and pain, provided by a nurse; (b) a 6-session structured psychosocial care protocol targeting depression and adjustment to illness, supplemented by informal (family) caregiver assessment and support, provided by a social worker or psychologist; and (c) brief weekly team meetings with the nurse, social worker/psychologist and a palliative care specialist, cardiologist, and primary care provider.
Period: Overall Study
Arm/Group | CASA | Psychospiritual
Started | 17 | 13
Completed | 16 | 7
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CASA | Psychospiritual | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [58 to 71] | 65 [58 to 66] | 63 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cohort Retention
Description: Cohort retention will be determined by examining the proportion of patients who complete the final study visit (at 3-month follow-up) over the total number of patients enrolled in the study (including deceased and lost-to-follow-up). Our goal is an 80% retention rate for this pilot study.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | CASA | Psychospiritual
Number analyzed (Participants) | 17 | 13
participants | 16 | 7

2. Secondary Outcome: Was Depression Addressed?
Description: The Patient Health Questionnaire-9 (PHQ-9) rates nine DSM-IV criteria of depression on a 0 (not at all) to 3 (nearly every day) scale. Scale range is 0-27, with depression severity scored: 0-4 (none), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), 20-27 (severe). The suicidal item is "thoughts that you would be better off dead, or of hurting yourself in some way?"
Time Frame: 3 months
Population: This analysis was only conducted in CASA participants
Measure: Number; unit: participants
Groups:
- CASA: A palliative symptom management and psychosocial care intervention named Collaborative Care to Alleviate Symptoms and Adjust to Illness that includes (a) evidence-based palliative symptom management of breathlessness, fatigue, and pain, provided by a nurse; (b) a 6-session structured psychosocial care protocol targeting depression and adjustment to illness, supplemented by informal (family) caregiver assessment and support, provided by a social worker or psychologist; and (c) brief weekly team meetings with the nurse, social worker/psychologist and a palliative care specialist, cardiologist, and primary care provider.
Arm/Group | CASA
Number analyzed (Participants) | 17
participants
  Baseline PHQ9 score >=10 | 4
  PHQ9 score >=10 addressed w/ treatment plan | 4
  Baseline PHQ9 suicidal item >=1 | 2
  PHQ9 suicidal item >=1 addressed w/ treatment plan | 2

3. Secondary Outcome: Participation Rates
Description: The investigators will use a CONSORT diagram to display participant flow, and determine how many of those who were approached enrolled in the trial.
Time Frame: 7 months
Population: The total population approached was 72 people. 31 consented to be randomized for a participate rate of 43%. Of these, one was a screen failure, and 17 and 13 were randomized to arm 1 and arm 2 respectively.
Measure: Number; unit: participants
Arm/Group | CASA | Psychospiritual
Number analyzed (Participants) | 72 | 72
participants | 17 | 13

4. Secondary Outcome: Adherence to the Study Protocol (CASA Arm Only)
Description: The investigators will calculate percentage adherence to pre-specified tasks on the intervention protocol, such as:
  * how often is depression addressed with a treatment plan?
  * how often are care team recommendations placed as orders in the medical record?
  * how often are orders completed?
Time Frame: 3 months
Population: A variety of process information was analyzed. Please see Bekelman DB et al, "Feasibility and acceptability of a collaborative care intervention to improve symptoms and quality of life in chronic heart failure: mixed methods pilot trial" Journal of Palliative Medicine 2014, PMID 14329424 for details.
Measure: Number; unit: %in arm severe target symptoms addressed
Arm/Group | CASA
Number analyzed (Participants) | 17
%in arm severe target symptoms addressed | 94

ADVERSE EVENTS:
Arm/Group | CASA | Psychospiritual
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No